CLINICAL TRIAL: NCT05427591
Title: Clinical and Microbiological Evaluation of the Chemo-mechanical Caries Removal Agent (BRIX3000®) in Primary Molars: A Randomized Controlled Clinical Trial.
Brief Title: Evaluation of the Chemo-mechanical Caries Removal Agent (BRIX3000®) in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Prof., King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Manal Maashi
Record Dates: First submitted 2019-06-25; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries
Keywords: BRIX3000; Carie-Care; Traditional surgical method; Microbiology; Pain; Primary molars
MeSH Terms: conditions — Dental Caries; Pain | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Experimental, two separate randomized controlled groups with split mouth design, following the "Consolidated Standards of Reporting Trials" (CONSORT,2010) statement. The final sample consisted of 60 children who met the inclusion criteria and had contralateral open occlusal carious lesions in their primary molars. They were randomly allocated to either group (1) or group (2). In group 1, 30 children with 60 primary molars underwent caries removal by the CMCR method "BRIX3000®" (the experimental group) on one molar (n = 30) and the traditional surgical method (the control group) on the contralateral molar (n = 30). In group 2, 30 children with 60 primary molars underwent caries removal by the CMCR method "Carie-CareTM" (the experimental group) on one molar (n = 30) and the traditional surgical method (the control group) on the contralateral molar (n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (1A) (Experimental): 30 children with 60 primary molars underwent caries removal by the CMCR method "BRIX3000®" (the experimental group) on one molar (n = 30).
  Interventions: Procedure: The chemomechanical caries removal agent "BRIX3000®" in group (1A)
- Group (1C) (Active Comparator): 30 children with 60 primary molars underwent caries removal by the traditional surgical method (the control group) on the contralateral molar (n = 30).
  Interventions: Procedure: The traditional surgical treatment in group (1C)
- Group (2B) (Experimental): 30 children with 60 primary molars underwent caries removal by the CMCR method "Carie-CareTM" " (the experimental group) on one molar (n = 30).
  Interventions: Procedure: The chemomechanical caries removal agent "Carie-CareTM" in group (2B)
- Group (2C) (Active Comparator): 30 children with 60 primary molars underwent caries removal by the traditional surgical method (the control group) on the contralateral molar (n = 30).
  Interventions: Procedure: The traditional surgical treatment in group (2C)

INTERVENTIONS:
Procedure: The chemomechanical caries removal agent "BRIX3000®" in group (1A) — In group(1A), the chemomechanical caries removal agent "BRIX3000®" was used for caries removal in primary molars.
  Arms: Group (1A)
Procedure: The traditional surgical treatment in group (1C) — In group(1C), the traditional surgical method (high-speed and low-speed air-rotors) was used for caries removal in primary molars.
  Arms: Group (1C)
Procedure: The chemomechanical caries removal agent "Carie-CareTM" in group (2B) — In group(2B), the chemomechanical caries removal agent "Carie-CareTM" was used for caries removal in primary molars.
  Arms: Group (2B)
Procedure: The traditional surgical treatment in group (2C) — In group(2C), the traditional surgical method (high-speed and low-speed air-rotors) was used for caries removal in primary molars.
  Arms: Group (2C)

SUMMARY:
Dental caries is one of the most prevalent chronic diseases in people worldwide. Traditional clinical treatment of dental decay has developed on the basis of the removal of carious tissues with high-speed handpieces and slow-rotating instruments, inducing pain, disturbing sounds, and vibrations. In addition, this method comprises the tooth structure by removing both "caries-affected dentin" and "caries-infected dentin". The use of the chemo-mechanical caries removal (CMCR) method is one of the main implementations of the minimal intervention dentistry idea accepted in the last ten years. It includes the selective removal of "caries-infected dentin" while preserving the healthy "caries-affected dentin" that has the ability to remineralize. The CMCR method differs from the traditional surgical method in that it selectively removes carious dentin. Therefore, it is less destructive and less painful, thereby promoting a positive attitude towards visiting dentists. A novel agent for the CMCR method named "BRIX3000®" by the laboratory Brix Medical Science has been released onto the dental market in 2016. It is a papain-based gel derived from latex and fruits of green papaya (Carica Papaya) that works as a chemical debridement with a unique technology called Encapsulating Buffer Emulsion (EPE). Investigations are required to evaluate and compare the outcomes of two CMCR agents, "BRIX3000®" and "Carie-CareTM," versus the traditional surgical methods. Therefore, the present study aims to perform a clinical and microbiological evaluation of caries removal using "BRIX3000®" and "Carie-CareTM" versus the traditional surgical methods in primary molars among children in Jeddah city, Saudi Arabia.

DETAILED DESCRIPTION:
Dental caries is one of the most prevalent chronic diseases in people worldwide. It results in localized dissolution and destruction of the calcified tooth tissues. The destruction of the dental structure does not occur as a result of a localized accumulation of bacteria, but rather as a result of an invasive and infectious process caused by the interaction of several interconnected factors. These factors make dental caries a great challenge for the dentist, as they seek an efficient means to control it. Carious dentin consists of two distinct layers: an outer "caries-infected dentin" and an inner "caries-affected". The "caries-affected" dentin is described as demineralized inter-tubular dentin, crystal deposition in dentinal tubules, and a lesser amount of destructed collagen matrix with no bacterial invasion. On the contrary, the "caries-infected" dentin displays deformation of the microstructure of the dentinal tubules and permanently damaged collagen fibers with significant penetration of the bacteria. Thus, the "caries-infected" dentin has to be removed only during caries removal. Traditional clinical treatment of dental decay has developed on the basis of the removal of carious tissues with high-speed handpieces and slow-rotating instruments, inducing pain, disturbing sounds, and vibrations. In addition, this method comprises the tooth structure by removing both "caries-affected dentin" and "caries-infected dentin". The concept of minimal intervention dentistry (e.g., air abrasion, laser, chemo-mechanical caries removal (CMCR) agents) includes the selective removal of caries-infected dentin while preserving the healthy caries-affected dentin that has the ability to remineralize. It is less destructive and less painful, thereby promoting a positive attitude towards visiting dentists among children. Brix Medical Science in 2016 released a new CMCR agent named "BRIX3000®". It is an enzymatic gel for non-traumatic caries removal known with exclusive technology as "Encapsulating Buffer Emulsion" (EPE) that is claimed to have superior characteristics for caries removal compared to previous products available in the dental market. There are a few studies present in the literature, most of them published in non-English language versions, evaluating the clinical and laboratory properties of "BRIX3000®". Therefore, investigations were required to evaluate and compare the outcomes of "BRIX3000®" versus the previous CMCR agent, "Carie-CareTM" and the traditional surgical methods. This study was carried out at King Abdulaziz Dental University Hospital (KADUH) and the Microbiology Research Laboratory in the Faculty of Pharmacy, King Abdulaziz University, Jeddah, Saudi Arabia to evaluate the efficacy, efficiency, and pain experienced by children with the use of the CMCR agents "BRIX3000®" and "Carie-CareTM" versus the traditional surgical method in primary molars. The study was approved by the "Research Ethics committee" at the Faculty of Dentistry, King Abdulaziz University (KAU) under approval number 107-06-19. Informed written consent will be signed by the parents/guardians of the children after explaining it to them. The study sample will be consisted of healthy and cooperative children aged 4 to 9 years old with bilateral open occlusal carious lesions in primary molars who will be seen as outpatients at KADUH's Department of Pediatric Dentistry from October 2019 to December 2020.The sample size was measured using G power analysis for calculating an estimated sample size. The final sample will be consisted of 60 children aged 4-9 years with 30 pairs of matched contralateral open occlusal carious lesions in primary molars meeting the inclusion criteria. They will be randomly allocated to either group (1) or group (2). In group 1, 30 children with 60 primary molars will be subjected to caries removal by the CMCR method "BRIX3000®" (the experimental group) on one molar (n = 30) and the traditional surgical method (the control group) on the contralateral molar (n = 30). In group 2, 30 children with 60 primary molars will be subjected to caries removal by the CMCR method "Carie-CareTM" (the experimental group) on one molar (n = 30) and the traditional surgical method (the control group) on the contralateral molar (n = 30). The block randomization method (a block of the two contralateral teeth) will be used to make sure that each side was treated evenly by both methods. The statistical assessment will be carried out using the Statistical Package for Social Sciences (SPSS, V.20, IBM, NY, USA). A significance level of 5% was utilized for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and cooperative patients of age group 4-9 years.
* Primary first/second molars with open occlusal carious lesion having moderated depth and clinically visible brownish color softened dentin.
* No clinical signs or symptoms of pulp degeneration, such as tenderness to percussion and history of sinus tracts or swelling. Intraoral periapical radiographs with lesions having radiolucency extending into, but only confined to dentin.

Exclusion Criteria:

* Patients with any major and minor systemic illness.
* Uncooperative patients that necessitate pharmacological dental treatment.
* Primary molars with mobile teeth, arrested caries, restored teeth, non-vital teeth, no carious lesion, presence of developmental defects and non-restorable teeth.
* Patients on any antibiotic regimen either on the day of treatment or for at least 2 weeks prior to the study.
* Patients allergic to Latex.
* Radiographic evidence of external or internal root resorption, furcal or periapical radiolucency.
* Primary molars with more than half of the root length resorbed.
* Children who did not attend and complete the second session of treatment.
* Not approving to sign the consent.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of caries removal | through study completion, an average of 1 year
  A change in the total viable count (TVC) of dentin samples taken during the dental treatment session is being assessed and presented as colony forming unit (CFU) per mL of sample.

SECONDARY OUTCOMES:
The efficiency of caries removal | through study completion, an average of 1 year
  The duration of the caries removal during the dental treatment session was recorded in minutes by a stopwatch.
The pain perception during caries removal | through study completion, an average of 1 year
  The Faces Pain Scale was used to evaluate the pain perception during the procedure of caries removal . The child was asked to choose a face (recorded with a score) matching the intensity of his or her pain experience during the procedure. The scores have a minimum value of 0 and a maximum value of 10. The higher the score, the more painful the procedure is.

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Elkhodary, D.Sc., Study Director — King Abdulaziz University; Najla'a M AL-Amoudi, D.Sc., Principal Investigator — King Abdulaziz University; Manal S Maashi, M.Sc., Study Chair — King Abdulaziz University
Locations (1):
- King Abdulaziz University, Dental University Hospital, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available within 18 months starting from 1st July 2019 for unlimited time.
Access Criteria: Public

REFERENCES:
- [Derived] Maashi M, Elkhodary H, Bamashmous N, Felemban O, Alamoudi N. Clinical performance of two chemomechanical caries removal agents in primary molars: a randomized controlled trial. Eur Arch Paediatr Dent. 2025 Aug;26(4):731-739. doi: 10.1007/s40368-025-01030-9. Epub 2025 Apr 9. PMID 40205159

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT05427591/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT05427591/ICF_001.pdf